CLINICAL TRIAL: NCT00922545
Title: Evaluation of a Combined Strategy Addressed to Practitioners and COPD Patients: Information Feed-back and Health Education, to Improve Clinical Control and Quality of Life
Brief Title: Evaluation of a Combined Strategy Addressed to Practitioners and Chronic Obstructive Pulmonary Disease (COPD) Patients to Improve Clinical Control and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Unitat de Suport a la Recerca de la Direcció d'Atenció Primària de Costa de Ponent (Unknown); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Carles Valero, Servei d'Atenció Primària Dreta.Institut Català de la Salut
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 550.62
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Quality of life; Primary health care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycophorins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Implementation of Clinical Practice Guidelines (GPC) and Health Education Program — Intervention: The program includes giving clinical results to the health care workers(doctor and nurse), from the medical records and interview. A training course (20h)that deals with aspects related to GPC, motivational interview and health education (tobacco, inhalers, alimentation, exercise and physiotherapy).

SUMMARY:
Main objective:

Evaluate the effectiveness of a combined strategy addressed to health care workers and patients, in relation to improving clinical control and patient's quality of life.It includes a feed-back about the health status of the patients, an education plan addressed to practitioners based in a CPG and in health education

DETAILED DESCRIPTION:
Method/design:

Design: Multicenter intervention study(before-after), quasi-experimental, prospective, with a control group and 12 month's follow-up

Setting: 21 primary Health Care Centres in Barcelona (Spain)

Sample: 801 patients (≥ 40 years old) with a register of COPD diagnostic,with one visit motivated by COPD during 2003 and that accept to participate at the study, after having read and signed the informed consent.

Intervention: The program includes giving clinical results to the health care workers(doctor and nurse), from the medical records and interview. A training course (20h)that deals with aspects related to GPC, motivational interview and health education (tobacco, inhalers, alimentation, exercise and physiotherapy).

Main variables: socio-demographic characteristics, quality of life, dyspnea, pharmacological treatment, exacerbations and hospital admissions, evaluation of inhalers technique, tobacco consumption, lifestyles and health resources used.

Measures: quality of life was evaluated with the Saint george's Respiratory Questionnaire (SGRQ) and dyspnea with the modified scale of the Medical Research Council (MRC). The variables are obtained at the beginning of the intervention and at the end (12 months after). Information about possible changes in lifestyle is gathered during the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged ≥40 years of age, recorded as having COPD, receiving attention in the PCC or at home, who have had at least one clinical visit for COPD management, and who provide written informed consent to participation in the study.

Exclusion Criteria:

* Patients who have any psychiatric disturbances, severe visual or auditory impairment that would impede compliance with the study protocol.
* Patients with asthma, tuberculosis or other chronic respiratory pathologies, or any end-stage disease, or not having access to a telephone.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2004-04; Primary Completion 2007-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life (Saint George's Respiratory Questionnaire (SGRQ) | Beginning of the intervention and at the end (12 months after)

SECONDARY OUTCOMES:
Dyspnea, exacerbations and hospital admissions | Beginning of the intervention and at the end (12 months after)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català de la Salut, Cornellà de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Valero C, Monteagudo M, Llagostera M, Bayona X, Granollers S, Acedo M, Ferro JJ, Rodriguez-Latre L, Almeda J, Munoz L; COPD Group of SAP Baix LLobregat Centre. Evaluation of a combined strategy directed towards health-care professionals and patients with chronic obstructive pulmonary disease (COPD): information and health education feedback for improving clinical monitoring and quality-of-life. BMC Public Health. 2009 Dec 1;9:442. doi: 10.1186/1471-2458-9-442. PMID 20128887